CLINICAL TRIAL: NCT03049241
Title: Neuromuscular Fatigue Aetiology Comparison Between Prepubertal Boys and Adults
Acronym: LENGTH-FATIG
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-304; 2016-A00827-44 (Other: 2016-A00827-44)
Record Dates: First submitted 2017-02-03; First posted 2017-02-10 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Neuromuscular Fatigue
Keywords: Children; Neuromuscular fatigue; Muscle group; Magnetic Nerve stimulation; Muscle length; Stiffness; prepubertal children; adults

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- knee extensors
  Interventions: Other: neuromuscular fatigue
- ankle plantar
  Interventions: Other: neuromuscular fatigue

INTERVENTIONS:
Other: neuromuscular fatigue — The main aim of the present protocol is to compare the effect of knee extensors and ankle plantarflexors length on the development and aetiology of neuromuscular fatigue, in children and adults

SUMMARY:
Potential factors involved in neuromuscular fatigue were classified into two categories: 1) central factors involving the central nervous system and neural pathways, and 2) peripheral factors occurring within the muscle beyond the neuromuscular junction. In adults, it has been shown that peripheral factors contribute to a large part of the fatigue induced by repeated maximal contractions. However in children, central factors could account for the development of fatigue to a greater extent. Force-generating capacity and musculotendinous stiffness could be two of the discriminatory factors accounting for the differences in the neuromuscular fatigue between children and adults.

Force production capacity and musculotendinous stiffness vary as function of muscle length. Naturally, they could differ depending on the muscle groups studied. The main aim of the present protocol is to compare the effect of knee extensors and ankle plantarflexors length on the development and aetiology of neuromuscular fatigue, in children and adults. The investigators formulated the hypotheses that at short muscle length force and low musculotendinous stiffness, differences in force between children and adults would be reduced. Thus neuromuscular fatigue development and aetiology would be similar between both groups. The results of the present protocol will allow to better understanding of the aetiology of neuromuscular fatigue in children and help improving training or rehabilitation programs.

DETAILED DESCRIPTION:
The study of neuromuscular fatigue in children is a recently topic in the field of sport sciences. Such knowledge could improve the efficiency and security of training and rehabilitation in healthy children and children with diseases like obesity.

The LENGTH-FATIG study will provide knowledge about the peripheral and central mechanisms of the neuromuscular fatigue in children and adults. Fatigue will test for different muscle groups (knee extensors and ankle plantar flexors) at different muscle lengths (short, optimal and long).

During high-intensity exercise, prepubertal children are more resistant to fatigue than adults. Contributions of the central and peripheral components to the development of neuromuscular fatigue are also different between both populations. The reduced children's fatigue coud be particularly related to a lower peripheral (i.e. muscular) fatigue. This might be attributed to the fact that prepubertal children rely more on oxidative than anaerobic metabolism than adults during fatiguing exercise. On the other hand, nervous factors could also explain differences in fatigue between children and adults. However, this topic is scarcely documented and still controversial. To our knowledge, no study has still compared the aetiology of central fatigue (supra-spinal vs. spinal) between children and adults. Only the voluntary activation level had been studied in children, conventionally used to assess central fatigue. But this factor doesn't differentiate spinal and supra-spinal contributions to neuromuscular fatigue development.

The LENGTH-FATIG research project is a physiological and observational study comparing two age groups (adults and children). Subjects will have to perform three randomized fatigue protocols at three muscle lengths (short, optimal and long) with the knee extensors and the ankle plantar flexors.

Data will be analyzed using LabChart 7.3 Pro software (ADInstrument, New South Wales, Australia) and Statistica 8.0 software (StatSoft, Inc.) and significance will be accepted at a two-sided alpha level of p<.05. The normality and homogeneity of the variables will be checked respectively from a Shapiro-Wilk test and a Barlett test.

If normality and homogeneity of the variables are verified, absolute values of variables (Force, EMG, NIRS, etc.) will be compared using three factors (age x muscle length x muscle group) analyses of variance (ANOVA) with repeated measures. If analyses reveal a significant effect of any factor or interaction of factors, post-hoc Newman-Keuls tests will be performed to determine differences between the different conditions.

If, on the contrary, normality and homogeneity of the variables are not verified, the effects of muscle length, muscle group and age will be evaluated using a Friedman test. If the tests show significant effects, comparisons of the different conditions will be performed using Mann-Whitney and Wilcoxon tests.

ELIGIBILITY:
Inclusion Criteria:

* Boys aged 8 to 11 years old, Tanner stages 1 to 3
* Male aged 18 to 35 years old
* Non-smoker
* Moderate physical activity level (< 4h/week)
* Covered by a social health insurance
* Consent form signed by participants and/or legal guardians.

Exclusion Criteria:

* Competitive training
* Cardiac or pulmonary diseases
* Epileptic seizures past history
* Magnetic field contraindication (including cardiac valve, pacemaker, prosthesis material, ferro-magnetic foreign body, cochlear implant and ocular prosthesis material.

Ages: 8 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: prepubertal boys and adults
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Maximal torque of knee extensors | once a week during six weeks.
ankle plantar flexors joint (in N.m) measured with a dynamometer. | once a week during six weeks.

SECONDARY OUTCOMES:
Doublet torque amplitude (100Hz, in N.m) evoked using magnetic nerve stimulation at rest | once a week during six weeks.
Muscular tissue oxygenation (in μmol.L-1) measured at skin surface by Near-infrared spectroscopy. | once a week during six weeks
Compound muscle action potential amplitude (i.e. M-wave ; in mV) evoked by supramaximal magnetic nerve stimulation and measured by surface Electromyography (EMG). | once a week during six weeks
High frequency doublet (100Hz)/low frequency doublet (10Hz) ratio | once a week during six weeks
fascicule length (mm) measured by B-mode real time ultrasound scanner. | once a week during six weeks
pennation angle (degree) measured by B-mode real time ultrasound scanner. | once a week during six weeks
Voluntary activation level (in %) assessed by using the twitch interpolation technique. | once a week during six weeks
EMG signal Root mean square of EMG signal during isometric maximal voluntary contractions. | once a week during six weeks
Hoffman reflex amplitude (i.e. H-reflex ; in mV) evoked by submaximal magnetic nerve stimulation measured by surface Electromyography (EMG). | once a week during six weeks
Cerebral tissue oxygenation (in μmol.L-1) measured at skin surface by Near-infrared spectroscopy | once a week during six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martine DUCLOS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France